CLINICAL TRIAL: NCT05485480
Title: Nociception Level During Opioid-sparing Anaesthesia Versus Conventional Opioid-based Anaesthesia: a Randomised Controlled Non-inferiority Trial
Brief Title: Nociception Level During Opioid-sparing Anaesthesia Versus Conventional Opioid-based Anaesthesia
Acronym: NOL_Basel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022-00283; qu20Bandschapp
Record Dates: First submitted 2022-07-20; First posted 2022-08-03 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Analgesia
Keywords: analgesia nociception; opioid-sparing anaesthesia; conventional opioid-based anaesthesia; Pain Monitoring Device (PMD-200); intraoperative nociceptive levels; Post operative nausea and vomiting (PONV)
MeSH Terms: conditions — Agnosia; Vomiting

STUDY DESIGN:
Intervention Model Description: Double blind, randomised controlled non-inferiority trial
Who Masked: Participant, Investigator
Masking Description: The patient and the investigator carrying out the nociception level measurement and the postoperative assessments will be blinded to the type of anaesthesia protocol that the patient is allocated to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Opioid-sparing: Lidocaine, Ketamine, Magnesium, Clonidine, Fentanyl, Remifentanil, Propofol (Experimental): Ketamine: started at 5mg/h; continued until 30min before end of surgery, then reduced to 1mg/h until discharge from recovery.
  Fentanyl: bolus of 50mcg before skin incision (in case of insufficient analgesia further boluses of 25mcg, upper limit is 100mcg).
  Lidocaine: bolus of 1.5mg/kg of ideal body weight (IBW),(maximum 100mg) at induction of anaesthesia, then continuous infusion of 1.5mg/kg IBW/h (maximum 100mg/h) until discharge from recovery.
  Magnesium: infusion of 2g/h for a maximum of 2h after induction of anaesthesia (maximum dose 4g). In case of bradycardia or hypotension, rate is reduced to 1g/h.
  Clonidine: bolus of 15mcg if needed. Maximum amount 150mcg. Remifentanil: started at time of induction of anaesthesia until end of surgery.
  Interventions: Drug: opioid-sparing group
- Conventional group: Fentanyl, Remifentanil, Propofol (Active Comparator): Control Intervention:
  Remifentanil: Remifentanil is given as a target controlled infusion using the Minto-model. It is started at the timepoint of induction of anaesthesia and given until the end of surgery.
  Fentanyl: 2mcg/kg i.v. is given at the time of induction of anaesthesia and another 1-2mcg/kg is given prior to incision. Further fentanyl boluses (1-2mcg/kg boluses) are given in case there seems to be insufficient analgesia.
  Interventions: Drug: conventional opioid-based group

INTERVENTIONS:
Drug: conventional opioid-based group — In addition to propofol as a hypnotic and rocuronium as a muscle relaxant, patients in the conventional opioid-based group will receive the following drugs: Remifentanil and Fentanyl
  Arms: Conventional group: Fentanyl, Remifentanil, Propofol
Drug: opioid-sparing group — In addition to propofol as a hypnotic and rocuronium as a muscle relaxant, patients in the opioid-sparing group will receive Ketamine, Fentanyl, Lidocaine, Magnesium, Clonidine, Remifentanil
  Arms: Opioid-sparing: Lidocaine, Ketamine, Magnesium, Clonidine, Fentanyl, Remifentanil, Propofol

SUMMARY:
The aim of this double blind, randomised controlled non-inferiority trial is to compare the antinociceptive efficiency of an opioid-sparing and a conventional opioid-based anaesthesia protocol with the help of the CEcertificated Pain Monitoring Device (PMD-200).

DETAILED DESCRIPTION:
Opioids have been an integral part of general anaesthesia. They are effective in preventing perception of noxious stimuli and ensure intraoperative haemodynamic stability. However, opioids are associated with a number of unwanted side effects (e.g. nausea and vomiting, sedation, ileus, respiratory depression, increased postoperative pain and morphine consumption and hyperalgesia). To minimise these side effects, there has been an interest in developing opioid-sparing anaesthesia protocols. Recently, analgesia nociception monitoring devices have become available. The aim of this double blind, randomised controlled non-inferiority trial is to compare the antinociceptive efficiency of an opioid-sparing and a conventional opioid-based anaesthesia protocol with the help of the CEcertificated Pain Monitoring Device (PMD-200). Patients scheduled to receive general surgical, gynaecological or urological laparoscopic surgery will be randomised into one of the two study groups. Study group A will be anaesthetised with an opioid-sparing protocol and study group B will be anaesthetised with a conventional opioid-based protocol. Intraoperative nociception will be evaluated with PMD-200. Postoperative visits will take place in recovery, 4-5h after surgery and then twice a day. In recovery, the amount of opioids and ketamine needed, pain, postoperative nausea and vomiting (PONV) and the time until the patient is fit for discharge according to the Aldrete score will be assessed. At the 4-5h postoperative visit, the amount of opioids and ketamine needed, maximum pain at rest and at mobilisation, incidence of PONV, mobilisation, micturition and sedation level will be assessed. At the twice daily follow up visits, amount of opioids and other analgesic drugs needed, pain at rest and at mobilisation, gastrointestinal function, quality of night's sleep, incidence of PONV, level of sedation and fitness for discharge home will be assessed. On day one after surgery, the perceived quality of recovery will be assessed with the QoR40 questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent as documented by signature
* Age older than 18 years
* Ability to give informed consent
* Undergoing scheduled general surgical, gynaecological or urological laparoscopic surgery
* American Society of Anesthesiology Score (ASA) status I, II, III

Exclusion Criteria:

* Inability to give informed consent
* ASA status IV and V
* Pregnant or breastfeeding women
* Allergy to one of the study drugs
* Urgent surgery
* Surgery with planned regional anaesthesia
* Outpatient surgery
* Atrioventricular block, intraventricular or sinoatrial block
* Atrial fibrillation
* Sinus bradycardia
* Cardiac insufficiency with a reduced left ventricular ejection fraction of below 40%
* Coronary artery disease
* Epilepsy
* Liver cirrhosis
* Chronic kidney disease (Clearance < 50ml/h)
* Chronic opioid therapy
* Chronic pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-17 (Actual); Primary Completion 2024-02-08 (Actual); Study Completion 2024-02-08 (Actual)

PRIMARY OUTCOMES:
Mean of the nociception level as measured by the PMD-200 | From the timepoint of skin incision until skin closure (within 1 day)
  The PMD-200 device consists of a finger probe which continuously assesses pulse rate, pulse rate variability, pulse wave amplitude, skin conductance level, skin conductance fluctuations, skin temperature, and finger motion. A value of 0 corresponds to no pain and a value of 100 to maximal pain. A value will be measured every minute from the timepoint of skin incision until skin closure.

SECONDARY OUTCOMES:
Change in Aldrete score | Every 15 minutes in recovery until patient discharge to the ward (within 1 day)
  Fitness for discharge to ward is checked every 15 minutes with the Aldrete score. The Aldrete score assigned a number of 0, 1, or 2 to 5 variables: activity, respiration, circulation, consciousness, and color. A score of 9 out of 10 is considered adequate for discharge from the recovery.
Amount of morphine needed | From the stay in recovery before discharge from the ward (average of 1 week)
  Amount of morphine needed
Amount of ketamine needed | From the stay in recovery before discharge from the ward (average of 1 week)
  Amount of ketamine needed
Change in pain score at rest by numeric rating scale | From the stay in recovery before discharge from the ward (average of 1 week)
  Change in pain score at rest by numeric rating scale (to assess pain severity using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable)
Change in pain score at movement by numeric rating scale | From the stay in recovery before discharge from the ward (average of 1 week)
  Change in pain score at movement by numeric rating scale (to assess pain severity using a 0-10 scale, with zero meaning "no pain" and 10 meaning "the worst pain imaginable)
Quality of night's sleep | From the first postoperative day until discharge from ward (average of 1 week)
  Quality of night's sleep assessed with a verbal numerical scale from 0 (very poor quality of sleep) to 10 (excellent quality of sleep)
Occurrence of nausea and vomiting | From the stay in recovery before discharge from the ward (average of 1 week)
  Occurrence of postoperative nausea and vomiting (PONV)
Change in level of sedation | At 4 hours and then twice daily until discharge from the ward (average of 1 week)
  Change in level of sedation
Perceived quality of recovery by QoR40 questionnaire | At the first postoperative day
  40-item questionnaire that provides a global score and subscores across five dimensions: patient support, comfort, emotions, physical independence, and pain
Time to return of gastrointestinal function | From the stay in recovery before discharge from the ward (average of 1 week)
  Time to return of gastrointestinal function as defined as the time from the end of surgery to the first passage of flatus and to the first bowel movement
Time to return of spontaneous micturition | From the stay in recovery before discharge from the ward (average of 1 week)
  Time to return of spontaneous micturition

CONTACTS AND LOCATIONS:
Overall Officials: Thierry Girard, Prof. Dr. med., Study Director — Department of Anaesthesiology, University Hospital Basel; Oliver Bandschapp, PD Dr. med., Principal Investigator — Department of Anaesthesiology, University Hospital Basel
Locations (1):
- Department of Anaesthesiology, University Hospital Basel, Basel, Switzerland